CLINICAL TRIAL: NCT02263430
Title: PINS Stimulator System for Deep Brain Stimulation in Huntington's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-007
Record Dates: First submitted 2014-09-28; First posted 2014-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Stimulation is on.
  Interventions: Device: Deep Brain Stimulation
- Placebo (Sham Comparator): Stimulation is off.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation
  Other Names: Rechargeable Neurostimulator

SUMMARY:
Deep Brain Stimulation (DBS) of the Globus pallidus internus(GPi) is useful in the treatment of different forms of chorea, including Huntington's disease (HD).

ELIGIBILITY:
Inclusion Criteria:

1. Subject clinically symptomatic and genetically confirmed Huntington Disease (number of CAG repeats>= 36)
2. Moderate stage of the disease (UHDRS motor>= 30)
3. Predominant movement disorder
4. Compliance of the patient, stable cognition during a 6 months phase prior to inclusion (Mattis Dementia Rating Scales（MDS）>/= 120)
5. Signed informed consent.

Exclusion Criteria:

1. Patients with hearing impairment;
2. Failures of important organs and in severe conditions;
3. Be reluctant or disabled to receive neuropsychological assessments;
4. Participate in other clinical trial;
5. Has a life expectancy of < 1 year.
6. The investigator and/or enrollment review committee, would preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Unified Huntington's Disease Rating Scale(UHDRS) | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University